CLINICAL TRIAL: NCT03061422
Title: Effect of Xylitol-Containing Chewing Gum With/Without Bicarbonate Versus Paraffin Pellet on Salivary pH in High Caries Risk Patients (A Randomized Clinical Trial)
Brief Title: Effect of Xylitol-Containing Chewing Gum With/Without Bicarbonate Versus Paraffin Pellet on Salivary pH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Howaida Fakhry Fouad, Resident of conservative departement , Faculty of Oral and Dental Medicine, Cairo university 2012, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEBC-CU-2017-02-14
Record Dates: First submitted 2017-02-19; First posted 2017-02-23 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Xylitol; Bicarbonates; Paraffin

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- xylitol chewing gum (Experimental): intervention
  Interventions: Other: Xylitol
- xylitol with bicarbonate chewing gum (Experimental): intervention
  Interventions: Other: xylitol with bicarbonate
- Paraffin pellet (Active Comparator): comparator
  Interventions: Other: paraffin

INTERVENTIONS:
Other: Xylitol — caries prevention chewing gum
  Arms: xylitol chewing gum
Other: xylitol with bicarbonate — caries prevention chewing gum
  Arms: xylitol with bicarbonate chewing gum
Other: paraffin — chewing gum
  Arms: Paraffin pellet

SUMMARY:
36 eligible participants will be randomly divided into three groups (n=12) according to the tested chewing gum (A), where (A1) represents participants exposed to xylitol chewing gum, (A2) represents participants exposed to bicarbonate and xylitol chewing gum and (A3) represents control group where participants are exposed to paraffin pellet chewing. The pH of saliva will be evaluated according to time in relation to the gum chewing (T) where (T0) represent the pH before chewing, (T1) represent 5 minutes after gum chewing at fixed time of the day (in the morning from 10 to 11 am).

Direct benefit of the research to the human volunteer:

It is important for high caries risk patients to decrease caries susceptibility as this will eventually decrease their dental treatments and subsequently the treatment cost.

Scientific value and social benefits:

This study will benefit the dentist as the main goal of a dentist is to prevent rather than cure. Also, it will decrease the restorative work carried out by dentist and save this time for educating more patients about caries prevention methods.

Expected risk to the human subjects:

Allergic reactions due to any of the components of the materials used which is rare to occur.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for the trial must comply with all of the following at randomization.

  1. Age range from 20-50 years
  2. High caries risk patients defined according to American Dental Association (ADA)
  3. Acidic baseline saliva pH
  4. Systematically healthy
  5. Not taking any medication interfering with saliva secretion
  6. Subjects who signed informed consent

Exclusion Criteria:

* (1) Subjects who wore orthodontic appliances or removable prosthesis (2) Subjects suffering from any medical or systematic disease (3) Smokers (4) Pregnant females (5) Allergy to any of chewing gum ingredients

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-03-03 (Estimated); Primary Completion 2017-10-01 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
Salivary pH change | an average of 1 year
  will be done by digital pH meter

CONTACTS AND LOCATIONS:
Locations (1):
- Howaida Fakhry Fouad, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ballal RK, Bhat SS, Ramdas SS, Ballal S. Effect of Chewing Bicarbonate-containing Sugar-free Gum on the Salivary pH: An in vivo Study. Int J Clin Pediatr Dent. 2016 Jan-Mar;9(1):35-8. doi: 10.5005/jp-journals-10005-1330. Epub 2016 Apr 22. PMID 27274153